CLINICAL TRIAL: NCT03568994
Title: A Trial of Atovaquone (Mepron®) Combined With Conventional Chemotherapy for de Novo Acute Myeloid Leukemia (AML) in Children, Adolescents, and Young Adults (ATACC AML)
Brief Title: Atovaquone (Mepron®) Combined With Conventional Chemotherapy for de Novo Acute Myeloid Leukemia (AML)
Acronym: ATACC AML
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Principal Investigator, Alexandra Stevens, M.D. Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-42691
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Atovaquone; Cytarabine; Daunorubicin; Etoposide; Gemtuzumab

STUDY DESIGN:
Intervention Model Description: Choice of Induction I regimen is at the treating physician's discretion (will be influenced based on drug availability)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADE 10+3+5 plus Atovaquone (AQ) (Experimental): Induction I ADE: cytarabine, daunorubicin, etoposide 10+3+5, atovaquone daily
- DA 3+10 with GO plus AQ (Experimental): Induction I DA: daunorubicin, cytarabine 3+10 with GO: gemtuzumab ozogamicin, atovaquone daily
  Interventions: Drug: Atovaquone; Drug: Cytarabine; Drug: Daunorubicin; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Atovaquone — Patients will receive standard of care MRC based Induction chemotherapy (such as ADE 10+3+5 with daily atovaquone dosing starting on day 6. In order to accommodate potential drug shortages modifications to ADE 10+3+5 that retain the MRC based induction backbone regimen of DA are allowed (see second Arm). These include but are not limited to substitution of etopophos for etoposide, exclusion of etoposide, use of CPX-351 (VYXEOS (daunorubicin and cytarabine) liposome) only, and daunorubicin and cytarabine (DA) + gemtuzumab ozogamicin (GO).
  Patients will be monitored for adherence to and tolerance of daily dosing of atovaquone. Peripheral blood (PB) and bone marrow plasma samples will be obtained to measure atovaquone concentrations.
  Other Names: Mepron
  Arms: DA 3+10 with GO plus AQ
Drug: Cytarabine — As part of routine Induction 1 chemotherapy (ADE 10+3+5)
  Arms: DA 3+10 with GO plus AQ
Drug: Daunorubicin — As part of routine Induction 1 chemotherapy (ADE 10+3+5)
  Arms: DA 3+10 with GO plus AQ
Drug: Etoposide — As part of routine Induction 1 chemotherapy (ADE 10+3+5)
Drug: Gemtuzumab Ozogamicin — As part of routine Induction 1 chemotherapy(DA 3+10 + GO)
  Arms: DA 3+10 with GO plus AQ

SUMMARY:
This study will test daily dosing of atovaquone at established pneumocystis jiroveci pneumonia (PJP) prophylaxis dosing in combination with standard induction chemotherapy for de novo AML. The primary objectives are to determine the frequency of omission of atovaquone doses due to standard induction chemotherapy toxicity, to quantify the steady-state plasma levels of atovaquone, and to determine the time to achievement of steady state atovaquone levels in this population.

DETAILED DESCRIPTION:
Standard cytotoxic chemotherapy is based on the Medical Research Council (MRC) backbone of cytarabine, and daunorubicin. This combination of chemotherapy is highly myelosuppressive and can lead to oral aversions, dietary intolerance, and gastrointestinal infections necessitating holding of oral drugs. Because of the toxicity of the best currently available therapy, new drugs that are considered for incorporation into existing treatment regimens will ideally have a tolerable side effect profile. This study will evaluate the tolerability of incorporating the orally bioavailable drug atovaquone in combination with standard cytotoxic induction chemotherapy for newly diagnosed pediatric AML patients. Therefore, quantifying the frequency with which atovaquone is held due to a side effect of therapy is crucial information to gather in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Children ≥1 month and children and young adults < 21 years of age
2. Diagnosis: Patients must be newly diagnosed with acute myelogenous leukemia

   2.1 Patients with previously untreated primary AML who meet the customary criteria for AML with ≥ 20% bone marrow blasts as set out in the 2008 World Health Organization (WHO) Myeloid Neoplasm Classification are eligible.

   Attempts to obtain bone marrow either by aspirate or biopsy must be made unless clinically prohibitive. In cases where it is clinically prohibitive, peripheral blood with an excess of 20% blasts and in which adequate flow cytometric and cytogenetics/Fluorescent in situ hybridization (FISH) testing is feasible can be substituted for the marrow exam at diagnosis

   2.2 Patients with < 20% bone marrow or peripheral blood blasts are eligible if they have:
   * A karyotypic abnormality characteristic of de novo AML (t(8;21)(q22;q22), inv(16)(p13q22) or t(16;16)(p13;q22) or 11q23 abnormalities,
   * The unequivocal presence of megakaryoblasts, or
   * Biopsy proven isolated myeloid sarcoma (myeloblastoma; chloroma, including leukemia cutis).
3. Pre-existing myelodysplastic syndrome:

   Patients with a history of myelodysplastic syndrome that has progressed to AML which meets the criteria above are eligible.
4. Therapy-related or secondary AML Patients with AML which is thought to be therapy related but meet the criteria above are eligible.
5. Prior Therapy:

   Prior therapy with hydroxyurea, all-trans retinoic acid (ATRA), corticosteroids (any route), and IT cytarabine given at diagnosis is allowed. Hydroxyurea and ATRA cannot be given concurrently with protocol therapy. There is no specific amount of time mandated between the last dose of hydroxyurea or ATRA and the start of protocol therapy.

   With the exception of infants who had previously received low dose cytarabine to control disease, patients who have previously received any other antileukemic therapy (i.e. chemotherapy or radiation therapy) are not eligible for this protocol.
6. Organ Function Requirement:

   Adequate Liver Function Defined as:
   * Direct Bilirubin ≤2x upper limit of normal (ULN) for age and institution (unless related to leukemic involvement), and
   * serum glutamate-pyruvate transaminase (SGPT) (ALT) ≤2.5x ULN for age and institution (unless it is related to leukemic involvement)
7. Ability to receive enteral medication:

Eligible patients should have no contraindication to enteral administration of medication (e.g. oral, Nasogastric (NG), G-tube, etc) as determined by the evaluating physician.

Exclusion Criteria:

1. Excluded Constitutional Conditions

   Patients with a history of any of the following constitutional conditions are not eligible:
   * Fanconi anemia
   * Shwachman syndrome
   * Any other known constitutional bone marrow failure syndrome
   * Patients with constitutional trisomy 21 or with constitutional mosaicism of trisomy 21 who are eligible to receive treatment for Down Syndrome (DS) related AML Note: Enrollment and initiation of therapy may occur pending results of clinically indicated studies to exclude these conditions. If a patient is found to have any of these conditions they should be removed from the study once results are received. Patients who are removed due to ineligibility after results are received will be replaced.
2. Other Excluded Conditions

   Patients with any of the following oncologic diagnoses are not eligible:
   * Any concurrent malignancy
   * Juvenile myelomonocytic leukemia (JMML)
   * Philadelphia chromosome positive AML
   * Biphenotypic or bilineal acute leukemia
   * Acute promyelocytic leukemia Note: Enrollment and initiation of therapy may occur pending results of clinically indicated studies to exclude these conditions. If a patient is found to have any of these conditions they should be removed from the study once results are received. Patients who are removed due to ineligibility after results are received will be replaced.
3. Prior receipt of anthracyclines Patients with treatment-related AML who have received more than 250mg/m2 of anthracyclines (in daunorubicin equivalents) are not eligible.
4. Known Allergy or Intolerance to Atovaquone Patients with a known allergy or intolerance to atovaquone are not eligible.
5. Enrollment on another ongoing treatment study Patients who are enrolled on a treatment study are not eligible
6. Pregnancy or Breast-Feeding 6.1 Female patients who are pregnant are ineligible since fetal toxicities and teratogenic effects have been noted for several of the study drugs.

   6.2 Lactating females are not eligible unless they have agreed not to breastfeed their infants.

   6.3 Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.
7. Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations | 5 weeks
  The investigators will determine plasma levels of atovaquone at the following time points: Day 6, 11, 13, 15, 18, 20, 22, 29 and on the day of the end of induction bone marrow (BM) assessment (generally around Day 36).
Dose Omission Frequency | 5 weeks
  To quantify the frequency of atovaquone doses omitted due to standard MRC related toxicity. Administration of doses of atovaquone will be monitored while the patient is hospitalized in the electronic medical record and abstracted to case report forms. Families will also be given a diary to complete.
Time to Achieve Steady State | 5 weeks
  Time to achieving steady state concentrations of atovaquone when given in combination with standard chemotherapy in children with de novo AML will be determined using stepwise tests of linear trend.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Stevens, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Baylor College of Medicine - Texas Childrens Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conneely SE, Stevens AM. Acute Myeloid Leukemia in Children: Emerging Paradigms in Genetics and New Approaches to Therapy. Curr Oncol Rep. 2021 Jan 13;23(2):16. doi: 10.1007/s11912-020-01009-3. PMID 33439382